CLINICAL TRIAL: NCT07405554
Title: Effect of Zinc Supplementation on Botulinum Toxin for Overactive Bladder: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Zinc Supplementation With Botulinum Toxin for Overactive Bladder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Ghazaleh Rostami Nia, Director of Research Division of Urogynecology, NorthShore University HealthSystem, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00000194
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Overactive Bladder (OAB)
Keywords: overactive bladder; botulinum toxin; zinc
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zinc + Phytase Group (Experimental): Participants will receive zinc + phytase capsules for five days prior to the scheduled procedure date.
  Interventions: Drug: Zinc Citrate Oral Capsule
- Placebo Group (Placebo Comparator): Participants will receive placebo capsules for five days prior to the scheduled procedure date.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zinc Citrate Oral Capsule — Zinc citrate 50mg combined with 7,500 phytase units in an oral capsule
  Arms: Zinc + Phytase Group
Drug: Placebo — Placebo oral capsule
  Arms: Placebo Group

SUMMARY:
This randomized, double-blind, placebo-controlled trial evaluates whether oral zinc plus phytase supplementation modifies clinical response to intradetrusor botulinum toxin injection in patients with overactive bladder. Participants will receive either zinc plus phytase supplementation or matching placebo for five days prior to intradetrusor botulinum toxin injection. Participants will be followed for six months after treatment to assess need for repeat botulinum toxin injection, urinary symptoms, and patient-reported outcomes related to overactive bladder.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

Intradetrusor botulinum toxin injection is an established treatment for overactive bladder (OAB) refractory to behavioral and pharmacologic therapy. However, duration of therapeutic effect varies among patients, and repeat injections are frequently required. Botulinum toxin activity depends on enzymatic cleavage of synaptic proteins involved in acetylcholine release, and zinc is a cofactor that may influence toxin activity. Phytase may enhance zinc bioavailability by improving intestinal absorption.

This study evaluates whether short-course oral zinc plus phytase supplementation administered prior to intradetrusor botulinum toxin injection alters clinical response to treatment.

STUDY OBJECTIVES

Primary Objective:

To determine whether oral zinc plus phytase supplementation prior to intradetrusor botulinum toxin injection reduces the proportion of patients requiring repeat intradetrusor botulinum toxin treatment within 6 months.

Secondary Objectives:

* To evaluate whether zinc plus phytase supplementation reduces urgency urinary incontinence episodes compared with placebo.
* To evaluate changes in overactive bladder symptom severity and patient-reported outcomes following treatment.
* To evaluate duration of clinical response following intradetrusor botulinum toxin injection.
* To evaluate safety and tolerability of short-course zinc plus phytase supplementation in this population.

STUDY DESIGN

This is a prospective, randomized, double-blind, placebo-controlled trial.

Participants with overactive bladder who are scheduled to undergo intradetrusor botulinum toxin injection as part of routine clinical care will be enrolled and randomized in a 1:1 ratio to receive either:

* Oral zinc plus phytase supplementation, or
* Matching placebo

Study medication will be administered for five days prior to the scheduled intradetrusor botulinum toxin injection.

Participants, investigators, and study personnel involved in outcome assessment will remain blinded to treatment assignment.

STUDY PROCEDURES

Participants will undergo intradetrusor botulinum toxin injection according to standard clinical practice.

Following injection, participants will complete remote follow-up assessments every four weeks for six months. Assessments will include:

* Bladder diaries
* Urinary symptom questionnaires
* Patient-reported outcome measures
* Assessment of retreatment status

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adult female at least 21 years old, with no plans to become pregnant during the course of the trial) and if of child-bearing potential, with a negative pregnancy test, and if sexually active, must be using medically acceptable contraception.
* ≥ 6 urgency urinary incontinence episodes on a 3-day baseline bladder diary, with these urge incontinence episodes representing greater than 50% of the total incontinent episodes recorded.
* Willing and able to complete all study related items and interviews.
* Refractory urgency urinary incontinence: defined as persistent symptoms despite at least one or more conservative treatments (e.g. supervised behavioral therapy, supervised physical therapy)
* Persistent symptoms despite the use of a minimum of two anticholinergics, or unable to tolerate medication due to side effects, or has a contraindication to taking anticholinergic/Beta 3 agonist medication.
* Currently not on an anticholinergic or antimuscarinic/Beta 3 agonist medication (e.g. oxybutynin, tolterodine, darifenacin, trospium chloride, solifenacin-succinate, fesoterodine and/or mirabegron) or be willing to stop medication for 3 weeks prior to completing baseline bladder diary and expected to remain off medications through duration of study.
* Demonstrates ability (or have caregiver demonstrate ability) to perform clean intermittent self-catheterization.
* Grossly neurologically normal on exam and no gross systemic neurologic conditions believed to affect urinary function.

Exclusion Criteria:

* Neurologic diseases such as multiple sclerosis, Parkinson Disease, CVA within 6 months prior to enrollment, myasthenia gravis, Charcot-Marie-Tooth disease, clinically significant peripheral neuropathy, and complete spinal cord injury.
* Untreated urinary tract infection (UTI).
* Any prior use of either study therapy for treatment of urinary urge incontinence (Botox A® or Interstim®).
* PVR >150 ml on 2 occasions within 6 months prior to enrollment (If the PVR value was obtained by ultrasound and was ≥150 ml, the PVR will be confirmed by catheterization which will be the gold standard).
* Current or prior bladder malignancy.
* Surgically altered detrusor muscle, such as augmentation cystoplasty.
* Subjects taking aminoglycosides.
* Currently pregnant or lactating.
* Allergy to lidocaine or bupivacaine.
* Prior pelvic radiation.
* Uninvestigated hematuria.

Ages: 21 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Need for repeat intradetrusor botulinum toxin injection at 6 months | 6 months
  Subjective patient report of need for repeat intradetrusor botulinum toxin injection at 6 months following index injection

SECONDARY OUTCOMES:
Urge urinary incontinence episodes assessed by 3-day Bladder Diaries | 6 months
  Mean number of urge urinary incontinence episodes based on 3-day bladder diaries
Urge urinary incontinence episodes assessed by PFDI-20 scores | 6 months
  Mean Pelvic Floor Distress Inventory-20 (PFDI-20) scores
Adverse events | 6 months
  Any adverse events that occur after intervention is administered

CONTACTS AND LOCATIONS:
Overall Officials: Ghazaleh Rostami Nia, MD, Principal Investigator — Endeavor Health
Locations (1):
- Endeavor Health, Skokie, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.